CLINICAL TRIAL: NCT03815396
Title: An Open-Label, Multicenter, Phase 1 Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Intravenous Doses of Inhibrx rhAAT-Fc (INBRX-101) in Adults With Alpha-1 Antitrypsin Deficiency (AATD)
Brief Title: Phase 1 Study to Assess the Safety, PK and PD of INBRX-101 in Adults With Alpha-1 Antitrypsin Deficiency
Acronym: rhAAT-Fc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inhibrx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ph1 INBRX-101
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Alpha-1 Antitrypsin Deficiency; AATD
Keywords: Alpha-1 antitrypsin deficiency; AATD; alpha-1 disease; AAT
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Single Ascending Dose (Experimental): INBRX-101 will be escalated in subjects with alpha-1 antitrypsin deficiency (AATD).
  Interventions: Drug: INBRX-101/rhAAT-Fc
- Part 2 Multiple Ascending Dose (Experimental): INBRX-101 will be escalated in subjects with alpha-1 antitrypsin deficiency (AATD).
  Interventions: Drug: INBRX-101/rhAAT-Fc

INTERVENTIONS:
Drug: INBRX-101/rhAAT-Fc — INBRX-101 is a recombinant human alpha-1 antitrypsin (AAT) Fc fusion protein (rhAAT-Fc).

SUMMARY:
This is an open-label, 2-part, dose-escalating, Phase 1 study of INBRX-101 (rhAAT-Fc). Part 1 will consist of single ascending dose (SAD) administration of INBRX-101 and Part 2 will consist of multiple ascending dose (MAD) administrations of INBRX-101. The planned dosing schedule is IV every 3 to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented alpha-1 antitrypsin (AAT) serum concentration <11 μM.
* Diagnosis of alpha-1 antitrypsin deficiency (AATD) with any allelic combination with exception of the null/null genotype.
* For subjects in Part 2 80 and 120 mg/kg cohorts ONLY: post-bronchodilator FEV1 of at least 40% of predicted normal value.
* For subjects in Part 2 80 and 120 mg/kg cohorts ONLY: subjects eligible for bronchoscopy per judgment of investigator.
* Nonsmoker for at least 6 months prior to study and must remain nonsmoking for the entire study duration.
* Adequate hepatic and renal function as defined per protocol.
* Willing to undergo current augmentation therapy washout (if applicable) and refrain from initiating augmentation therapy, other investigational drug trials for AATD, therapy with IV immunoglobulins or monoclonal antibodies during the entire study, including follow-up.

Exclusion Criteria:

* Known or suspected allergy to components of INBRX-101 (AAT or human IgG) or pdAAT.
* Participation in any investigational drug trial within 30 days prior to this trial, or subjects receiving IV immunoglobulins or monoclonal antibodies within 30 days prior to this trial.
* History of and/or on the waiting list for lung or liver transplant, lobectomy, or lung volume reduction surgery.
* Acute respiratory tract infection or COPD exacerbation that required antibiotic treatment and/or increase in systemic steroid dosage within the 4 weeks prior to screening. Subjects are permitted to continue to receive steroids if the investigator judges the subject to have a history of stable dosing.
* Subjects with ongoing or history of unstable cor pulmonale.
* Infection with hepatitis A, B, or C or human immunodeficiency virus (HIV).
* Active autoimmune disease or documented history of autoimmune disease that 1) required systemic steroids or immune-suppressive medications and 2) tested positive for auto-antibodies. Exception: Endocrinopathies managed with hormone replacement therapy (HRT).
* Current substance and/or alcohol abuse with protocol defined exceptions.
* Current narcotics abuse with protocol defined exceptions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events of INBRX-101 | Up to 7 months
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03.
Severity of adverse events of INBRX-101 | Up to 7 months
  Severity of adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03.

SECONDARY OUTCOMES:
Area under the serum concentration time curve (AUC) of INBRX-101 | Up to 7 months
  Area under the serum concentration time curve (AUC) of INBRX-101 will be determined.
Maximum observed serum concentration (Cmax) of INBRX-101 | Up to 7 months
  Maximum observed serum concentration (Cmax) of INBRX-101 will be determined.
Trough observed serum concentration (Ctrough) of INBRX-101 | Up to 7 months
  Trough observed serum concentration (Cmax) of INBRX-101 will be determined.
Time to Cmax (Tmax) of INBRX-101 | Up to 7 months
  Time to Cmax (Tmax) of INBRX-101 will be determined.
Half-life (T1/2) of INBRX-101 | Up to 7 months
  Half-life of INBRX-101 will be determined.
Immunogenicity of INBRX-101 | Up to 7 months
  Frequency and consequences of anti-drug antibodies (ADA) against INBRX-101 will be determined.
Distribution of INBRX-101 in Bronchoalveolar Lavage Fluid (BALF) | Up to 7 months
  The concentration of INBRX-101 in bronchoalveolar lavage fluid (BALF) be determined.
Functional concentration of INBRX-101 in serum and BALF | Up to 7 months
  The functional concentration of INBRX-101 in serum and BALF will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Andrianov, MD, Study Director — Inhibrx Biosciences, Inc
Locations (10):
- United States (5):
  - UC Davis School of Medicine, Sacramento, California
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Hannibal Clinic, Hannibal, Missouri
- New Zealand (3):
  - The New Zealand Respiratory and Sleep Institute, Auckland
  - Christchurch Clinical Studies Trust Ltd, Christchurch
  - Waikato Respiratory and Gastro Research Unit, Hamilton
- United Kingdom (2):
  - University of Cambridge, Cambridge, East of England
  - University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No